CLINICAL TRIAL: NCT06554236
Title: The Influence of an Orthopaedic Manual Physical Therapy Approach and Sensory Training on Somatoperception in Patients with Chronic Low Back Pain
Brief Title: The Influence of an Orthopaedic Manual Physical Therapy and Sensory Training on Somatoperception in Patients with Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brooke Barletta, Principal Investigator, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.2024.071d
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain
Keywords: two-point discrimination; physical therapy; somatoperception; tactile acuity
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: quasi-experimental, one-group repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic low back pain (Experimental): 18-64 years with low back pain duration > 3 months.
  Interventions: Other: physical therapy and sensory training

INTERVENTIONS:
Other: physical therapy and sensory training — Physical therapy standard of care and 5 minutes of sensory training.

SUMMARY:
Individuals with chronic low back pain and other chronic pain conditions have been shown to have altered somatosensory, the ability to sense input to the tissue, which is processed in the primary somatosensory cortex or S1. Two-point discrimination is currently the best clinical tool utilized to assess an individual's ability to sense touch. This study will assess TPD changes after a course of standard physical therapy care with the addition of sensory training.

ELIGIBILITY:
Inclusion Criteria:

* DEERS eligible
* 18 to 64 years old
* Low back pain > 3 months
* Numeric Pain Rating Scale minimal pain rating of 3/10 in the last seven days
* Must be able to commit to 6-10 treatment sessions over a period of at least 6-we

Exclusion Criteria:

* History of spinal surgery
* History of spinal injections or nerve ablations in the past year
* History of traumatic brain injury (TBI)
* History of cerebral vascular accident (CVA)
* Currently pregnant
* Active cancer
* Symptoms below the knee
* Non-MSK condition contributing to low back pain
* Chronic Pain Conditions to include Chronic Regional Pain Syndrome and Fibromyalgia
* Autoimmune Diseases (to include Ankylosing Spondylitis, Lupus, Rheumatoid Arthritis)
* Currently under litigation related to low back pain
* Currently going through Medical Evaluation Board (MEB)
* Retiring or separating from the military within a year
* Currently receiving physical therapy for low back pain

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Tactile acuity as measured by two-point discrimation | Performed at baseline visit, 4th week of treatment, and at final visit (8 +/- 2 weeks).
  measured using a Caroline 2-point discriminator tool. TPD is the most widely accepted objective measurement of tactile acuity in the clinical setting

SECONDARY OUTCOMES:
Pain as measured by numeric pain rating scale | Performed at baseline, 4th week of treatment, and final visit (8 +/- 2 weeks).
  The NPRS is an 11-point numerical pain rating scale used to measure pain. Patients rate pain ranging between 0 (no pain) and 10 (worst pain imaginable)
Low back perception | Performed at baseline, 4th week of treatment, and final visit (8 +/- 2 weeks).
  measured using the Freemont Back Awareness Questionnaire (FreBAQ), a multi-item, self-report questionnaire designed to quantify distorted perception of the back in people with CLBP
Tactile Localization Accuracy | Performed at baseline, 4th week of treatment, and final visit (8 +/- 2 weeks).
  measured by the number of correct responses out of 9 attempts for stimulation of the 9-grid chart
Function | Performed at baseline, 4th week of treatment, and final visit (8 +/- 2 weeks).
  measured by the Oswestry Disability Index (ODI), 10 patient-completed questions in which the response options are presented as 6-point Likert scales. Scores range from 0% (no disability) to 100% (most severe disability

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Barletta, Principal Investigator — Brooke AMC

IPD SHARING:
Plan to Share IPD: Yes
Requests for deidentified data will be considered on a case by case basis.
Supporting Information: Study Protocol
Time Frame: Requests for deidentified data will be considered on a case by case basis.
Access Criteria: Requests for deidentified data will be considered on a case by case basis.
URL: https://bamc.tricare.mil/